CLINICAL TRIAL: NCT07123220
Title: Identification of Prognostic Factors for Fatigue in Patients With Systemic Lupus Erythematosus. A Multicenter Cross-sectional Cohort Study
Brief Title: Prognostic Factors for Fatigue in Patients With Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, Investigación en Hemofilia y Fisioterapia
Other Study IDs: Lup-Obs
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus; Fatigue; Anxiety; Quality of life; Physical activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients who meet the selection criteria will be informed of the characteristics, objectives, and risks of the evaluation. They will be provided with patient information and informed consent documents. After confirming that they do not meet any of the exclusion criteria, the dependent and confounding variables of the study will be evaluated.
  The assessment will be carried out using self-questionnaires that will be sent online to the various associations of patients with systemic lupus erythematosus that are part of the Spanish Lupus Federation. All questionnaire assessments will be carried out by the same physical therapist, following the same assessment protocol.

SUMMARY:
Introduction: Fatigue is a well-established symptom in systemic lupus erythematosus. Depression and anxiety can develop at different stages of systemic lupus erythematosus and their severity can range from mild symptoms to more serious disorders. Patients with systemic lupus erythematosus may consider fatigue to be a symptom that is more severe than pain, depression, or anxiety.

Objectives: To describe fatigue in patients with systemic lupus erythematosus and identify the best predictive model for fatigue in these patients.

Methods: Multicenter cross-sectional cohort studies. Eighty-eight patients with systemic lupus erythematosus from different regions of Spain will be included in the studies. The primary variable will be fatigue (Fatigue Assessment Scale), with anxiety (State-Trait Anxiety Inventory) as the dependent variable. The secondary variables will be perceived quality of life (Lupus Quality of Life and 36-Item Short Form Survey Instrument), level of physical activity (International Physical Activity Questionnaire), and the main clinical, sociodemographic, and anthropometric variables.

Expected results: To describe fatigue in patients with systemic lupus erythematosus, as well as the predictive model for fatigue in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with systemic lupus erythematosus.
* Over 18 years of age.
* Who have not had any flare-ups in the last 6 months.
* Who sign the informed consent form.

Exclusion Criteria:

* Patients with neurological or cognitive impairments that prevent them from understanding the questionnaires and physical tests.
* Patients who are receiving an intervention (physiotherapy or orthopedic) at the time of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus. A total of 88 patients are expected to be included in this project.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of fatigue at baseline | Baseline
  Fatigue will be assessed using the Fatigue Assessment Scale. This tool provides information on the physical and psychological aspects of fatigue. This scale is highly reliable. This self-reported questionnaire consists of 10 items with a 5-point Likert response scale. Five items reflect the physical component and five reflect the psychological component. The score range of the scale is 10-50 (the higher the score, the greater the degree of fatigue).

SECONDARY OUTCOMES:
Assessment of anxiety symptoms at baseline | Baseline
  The State-Trait Anxiety Inventory will be used to measure the presence and severity of anxiety symptoms in patients with systemic lupus erythematosus. There are two subscales within this measure: state and trait. The state anxiety scale assesses the current state of anxiety, while the trait anxiety scale assesses relatively stable aspects of the propensity for anxiety. This scale has 40 items, 20 assigned to each of the subscales, with a range of 1 to 4 points (the higher the score, the higher the level of anxiety).
Assessment of quality of life at baseline | Baseline
  Quality of life in patients with systemic lupus erythematosus will be measured using the Spanish version of the Lupus Quality of Life (LupusQoL) questionnaire. This questionnaire consists of 34 items in 8 domains (physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden on others). The questionnaire scores range from 0 (worst quality of life) to 100 (best quality of life).
Assessment of health-related quality of life at baseline | Baseline
  The Spanish version of the Short Form-36 Health Survey (SF-36) questionnaire will be used to measure health-related quality of life. It consists of 36 items that investigate eight dimensions (physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health, including a health transition item). The score ranges from 0 to 100 (better perception of quality of life).
Assessment of physical activity level at baseline | Baseline
  Physical activity level will be assessed using the International Physical Activity Questionnaire (IPAQ). This tool consists of seven questions that inquire about the frequency, duration, and intensity of physical activity performed in the last week. It also assesses the time spent walking and sitting. The results are classified into three categories: low, moderate, and high activity, identifying whether individuals meet the WHO activity recommendations. The unit of measurement is the metabolic equivalent of task (METS), where a higher number of METS indicates greater physical activity.
Assessment of lupus activity index at baseline | Baseline
  The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a widely used tool in the evaluation of systemic lupus erythematosus. This global index assesses disease activity over the last 10 days and consists of 24 items that collect specific manifestations in 9 organs or systems. The SLEDAI score ranges from 0 to 105, with higher scores indicating greater disease activity.
Assessment of cumulative damage in lupus at baseline | Baseline
  The assessment of cumulative damage in patients with systemic lupus erythematosus will be performed using the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR). The tool includes 12 organ systems and measures irreversible damage from the onset of the disease, regardless of its activity, adverse effects due to treatment, or comorbidities. For damage to be considered, it must have been present for at least six months, thus avoiding confusion with active inflammatory processes. The total index score ranges from 0 to 46, with a higher score indicating a greater degree of cumulative damage.

OTHER OUTCOMES:
Assessment of the sociodemographic variable age at baseline | Baseline
  The sociodemographic variable 'age' will be measured in full months from the patient's date of birth to the date of assessment.
Assessment of the sociodemographic variable marital status at baseline | Baseline
  The sociodemographic variable marital status will be measured using 4 response options (qualitative variable): single / married / divorced / widowed.
Assessment of the sociodemographic variable sex at baseline | Baseline
  The sociodemographic variable sex will be measured using a dichotomous variable (Male/Female)
Assessment of the sociodemographic variable educational level at baseline | Baseline
  The sociodemographic variable educational level will be measured using 4 response options (qualitative variable): primary education / secondary education / university education / postgraduate education.
Assessment of the sociodemographic variable employment status at baseline | Baseline
  The sociodemographic variable employment status will be measured using 4 response options (qualitative variable): self-employed / employed by others / unemployed / disability-retirement.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Almería, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No